CLINICAL TRIAL: NCT00345683
Title: Single-blind, Randomized, Controlled, Multinational Study for the Evaluation of Safety of GSK Biologicals' Hib-MenCY-TT Vaccine Compared to Monovalent Hib Control Vaccine in Healthy Infants at 2, 4, 6, and 12 to 15 Months of Age.
Brief Title: Safety of Hib-MenCY-TT Vaccine Versus Licensed Hib Conjugate Vaccine, Given at 12 to 15 Months of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 105988
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: H. influenzae type B vaccine; Infants; Neisseria meningitidis; Vaccines, conjugate; Meningococcal vaccines; Prophylaxis; Comparative study; Safety; Humans
MeSH Terms: conditions — Haemophilus Infections | interventions — Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine; Heptavalent Pneumococcal Conjugate Vaccine; Measles-Mumps-Rubella Vaccine; Rubella Vaccine; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- Menhibrix Group (Experimental): Subjects received 3 doses of Menhibrix vaccine (at 2, 4 and 6 months of age, study Months 0, 2 and 4), co-administered with Pediarix/Infanrix penta as a primary vaccination course in the study NCT00345579 and a fourth dose of Menhibrix vaccine at 12-15 months of age in this study (study Month 10-13). Menhibrix was administered intramuscularly in the upper right thigh and co-administered Pediarix/Infanrix penta vaccine was injected intramuscularly in the upper left thigh.
  Interventions: Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine combined (792014); Biological: Prevnar; Biological: M-M-R II; Biological: Varivax
- ActHIB Group (Active Comparator): Subjects received 3 doses of ActHIB vaccine (at 2, 4 and 6 months of age, study Months 0, 2 and 4), co-administered with Pediarix/Infanrix penta as a primary vaccination course in the study NCT00345579 and 1 dose of PedvaxHib vaccine as a booster at 12-15 months of age in this study (study Month 10-13). ActHIB and PedvaxHib vaccines were administered intramuscularly in the upper right thigh and co-administered Pediarix/Infanrix penta vaccine was injected intramuscularly in the upper left thigh.
  Interventions: Biological: PedvaxHIB; Biological: Prevnar; Biological: M-M-R II; Biological: Varivax

INTERVENTIONS:
Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine combined (792014) — Booster dose by intramuscular injection
  Arms: Menhibrix Group
Biological: PedvaxHIB — Booster dose by intramuscular injection
  Other Names: Monovalent Hib conjugate vaccine.
  Arms: ActHIB Group
Biological: Prevnar — Booster dose by intramuscular injection
Biological: M-M-R II — Single dose by subcutaneous injection
  Other Names: Measles; mumps and rubella vaccine.
Biological: Varivax — Single dose by subcutaneous injection
  Other Names: Varicella vaccine

SUMMARY:
The booster phase of the study will evaluate the safety of Hib-MenCY-TT vaccine compared to a control group receiving licensed Hib conjugate vaccine at 12 to 15 months of age.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00345579).

No new recruitment will take place during this booster phase of the study. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Hib-MenCY-TT = GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine.

The study will be conducted in a single blind manner up to 30 days after administration of the booster dose; the extended safety follow-up after the booster dose will be conducted in an unblinded manner.

All subjects will receive Prevnar, M-M-R II and Varivax as study vaccines, preferencially co-administered with the booster dose of Hib-MenCY-TT/PedvaxHIB.

Note: This protocol posting deals with the objectives & outcome measures for the booster phase of the study. The objectives & outcome measures for the primary phase are presented in a separate protocol posting (NCT00345579)

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in the primary study (NCT00345579) are eligible for participating in the booster study

Exclusion Criteria:

Subjects should not be administered M-M-R II and Varivax if any of these criteria apply:

* History of measles, mumps, rubella or varicella.
* Previous vaccination against measles, mumps, rubella or varicella.
* Hypersensitivity to any component of the vaccines, including gelatin or neomycin.
* Patients receiving immunosuppressive therapy.
* Individuals with blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Individuals with primary and acquired immunodeficiency states.
* Individuals with a family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* Individuals with active tuberculosis.
* Acute disease at time of booster vaccination

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4021 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (48):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Madera, California
  - GSK Investigational Site, Slinas, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Waukee, Iowa
  - GSK Investigational Site, West Desmoines, Iowa
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Nies, Michigan
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, New Hartford, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Boardman, Ohio
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, North Canton, Ohio
  - GSK Investigational Site, South Euclid, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wexford, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Pleasant Gorve, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin
- GSK Investigational Site, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Rinderknecht S, Bryant K, Nolan T, Pavia-Ruz N, Doniz CA, Weber MA, Cohen C, Aris E, Mesaros N, Miller JM. The safety profile of Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine (HibMenCY). Hum Vaccin Immunother. 2012 Mar;8(3):304-11. doi: 10.4161/hv.18752. Epub 2012 Feb 13. PMID 22327493
- See also: Primary Study — http://www.clinicaltrials.gov/ct/show/NCT00345579
- Available data/document: Informed Consent Form: 105988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 105988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This summary presents results for the booster/fourth dose vaccination phase up to the end of the 6-month safety follow-up. Subjects received 3-vaccine doses in the study NCT00345579 and were followed up to, but excluding, the fourth dose vaccination. This study begins 10 months after the first vaccination in the primary phase.
Pre-assignment Details: Of the 4021 subjects enrolled, 4020 received a booster vaccination and 3986 completed the booster phase (2985 in the Menhibrix Group and 1001 in the ActHIB Group)
Period: Overall Study
Arm/Group | Menhibrix Group | ActHIB Group
Started | 3010 | 1010
Completed | 2985 | 1001
Not Completed | 25 | 9
Not completed — Lost to Follow-up | 19 | 7
Not completed — Other | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menhibrix Group | ActHIB Group | Total
Number analyzed (Participants) | 3010 | 1010 | 4020
Age, Continuous [Mean (Standard Deviation); unit: Days] | 12.1 (0.34) | 12.1 (0.33) | 12.1 (0.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1450 | 505 | 1955
  Male | 1560 | 505 | 2065

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: From fourth dose up to Day 30 after fourth dose vaccination (from study Month 10-13 up to study Month 11-14)
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 12 | 1

2. Primary Outcome: Number of Subjects Reporting New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From fourth dose up to Day 30 after fourth dose vaccination (from study Month 10-13 up to study Month 11-14)
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 12 | 6

3. Primary Outcome: Number of Subjects Reporting Rash
Description: Rash assessed was hives, idiopathic thrombocytopenic purpura, petechiae
Time Frame: From fourth dose up to Day 30 after fourth dose vaccination (from study Month 10-13 up to study Month 11-14)
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 123 | 41

4. Primary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER) Visits
Time Frame: From fourth dose up to Day 30 after fourth dose vaccination (from study Month 10-13 up to study Month 11-14)
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 29 | 16

5. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 72 | 18

6. Primary Outcome: Number of Subjects With New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: as for outcome 5
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 50 | 18

7. Primary Outcome: Number of Subjects With Rash
Description: Rash assessed was hives, idiopathic thrombocytopenic purpura, petechiae
Time Frame: as for outcome 5
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 227 | 82

8. Primary Outcome: Number of Subjects With Adverse Events Resulting in Emergency Room (ER) Visits
Time Frame: as for outcome 5
Population: The Fourth dose Total Vaccinated cohort included all subjects who received the fourth study dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3010 | 1010
Subjects | 129 | 48

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Description: Only information about specific categories of AEs (SAEs, NOCIs, rash and AEs resulting in ER visits) were collected in this study. Data for unsolicited AEs and solicited symptoms were not collected.
Arm/Group | Menhibrix Group | ActHIB Group
Serious Adverse Events (participants affected / at risk) | 72/3010 | 18/1010
Other Adverse Events (participants affected / at risk) | 0/3010 | 0/1010
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menhibrix Group (N=3010) | ActHIB Group (N=1010)
Gastroenteritis (Infections and infestations) | 28 | 7 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Dehydration (Metabolism and nutrition disorders) | 6 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Bronchiolitis (Infections and infestations) | 8 | 3 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Staphylococcal infection (Infections and infestations) | 2 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Abscess (Infections and infestations) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Febrile convulsion (Nervous system disorders) | 6 | 2 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Head injury (Injury, poisoning and procedural complications) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Otitis media (Infections and infestations) | 1 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Pyrexia (General disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Pneumonia (Infections and infestations) | 3 | 2 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Croup infectious (Infections and infestations) | 0 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Ataxia (Nervous system disorders) | 1 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Bronchopneumonia (Infections and infestations) | 2 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Influenza (Infections and infestations) | 2 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Pneumonia bacterial (Infections and infestations) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Upper respiratory tract infection (Infections and infestations) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Erysipelas (Infections and infestations) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Folliculitis (Infections and infestations) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Subcutaneous abscess (Infections and infestations) | 0 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)
Tracheitis (Infections and infestations) | 0 | 1 — From fourth dose through the end of the 6-month safety follow-up of the fourth dose phase (from study Month 10-13 up to study Month 16-19)

LIMITATIONS AND CAVEATS:
Only information about specific categories of AEs (SAEs, NOCIs, rash and AEs resulting in ER visits) were collected in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.